CLINICAL TRIAL: NCT00338520
Title: Hyperphenylalaninemia in Cerebral Malaria
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Hubert Kairuki Memorial University (Other); Duke University (Other); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14617; 05-0116
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Cerebral malaria, phenylalanine, Tanzania
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Cerebral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, CSF, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Controls (HC): Healthy control children will be enrolled from out-patient well-baby visits.
- Uncomplicated Malaria (UM): Febrile children admitted to the hospital with Plasmodium falciparum parasitemia, no other cause of fever identified, no evidence of severe malaria (as listed in Study Protocol, Section 5.2 under exclusion criteria for UM), and no co-infection with other malaria species will be enrolled in the UM group.
- Cerebral Malaria (CM): Comatose children admitted to the hospitals will be evaluated by the house physician and/or member of the study team. If lumbar puncture is obtained, the parent or guardian will be approached for permission to enroll the child into the study. Parasitemic children with no other cause of coma identified will included in the CM group.
- Non-malaria CNS disease (NMC): Children without parasitemia and diagnosed with a non-malaria cause of coma or CNS disease will be enrolled in the non-malaria CNS disease group.

SUMMARY:
The purpose of this study is to see if children, who develop coma from malaria, are not making enough of a vitamin-like chemical, tetrahydrobiopterin (BH4), which is required for the brain to function normally. This information may help to identify new ways to treat malaria in the future. Study participants will include 512 children, ages 6 months to 6 years. Participants will be placed into one of 4 groups: well children; children with mild malaria; children without malaria, but with a medical problem involving the brain that requires a lumbar puncture for diagnosis (a procedure in which a needle is placed into an area surrounding the spinal cord and a sample of cerebral spinal fluid is removed); and children with a severe form of malaria affecting the brain called cerebral malaria. Study procedures will include blood samples, urine samples and lumbar puncture, only if necessary for diagnosis as part of standard practice procedures. Participants will be involved in study related procedures for up to 3 weeks.

DETAILED DESCRIPTION:
The mortality in severe malaria remains between 12-30% despite antimalarial therapy. The overwhelming majority of deaths from malaria occur in children in impoverished countries of the world with cerebral malaria (CM) and metabolic acidosis as the most important negative prognostic indicators. CM is a serious complication of falciparum malaria. It is characterized by fever, coma (not attributable to hypoglycemia), seizures (not attributable to febrile seizures) and abnormalities of muscle tone (rigidity, hypotonia) and body posture (decerebrate, decorticate, opisthotonic posturing). This observational prospective cohort study will enroll 512 Tanzanian children, 6 months to 6 years old, admitted to the hospital with CM (Group 1) as defined by World Health Organization criteria and uncomplicated malaria (UM-Group 2). Healthy children who are not acutely ill (healthy control, HC-Group 4) and children with coma and/or central nervous system (CNS) illness not attributed to malaria (NMC-Group 3) will serve as controls. Children will be recruited from 2 hospitals in Dar es Salaam, Amana Hospital in the Ilala District (AHID) and Mwananyamala Hospital (MDH)in the Kinondoni District. Children presenting to AHID or MDH, who are diagnosed with CM or a non-malarial CNS condition will be transferred by ambulance to the Clinical Research Unit (CRU) at Hubert Kairuki Memorial University (HKMU). Before transfer the child will be stabilized and treatment will be initiated. A lumbar puncture will be performed. Transfer to the HKMU-CRU will take place only with the parent(s)/guardian(s) permission and the parent(s) and/or guardian(s) will be transferred to HKMU with the child. Comatose children admitted to the hospitals will be evaluated by the house physician and/or member of the study team. Febrile children admitted to the hospital with high level Plasmodium falciparum parasitemia, no other cause of fever identified, nor evidence of severe malaria and no co-infection with other malaria species will be enrolled in the UM group. Health control children will be enrolled from outpatient well-baby clinics at AHID and MDH. All ill (groups II, III, IV)children will have complete blood picture, urinalysis, blood culture, and a blood smear for malaria. Lumbar puncture will be performed for diagnosis of meningitis or hemorrhage (in groups I and III) if there are no contraindications (e.g. papilledema or focal neurological signs suggesting a CNS mass lesion). Children will be treated according to Tanzanian standards based on the initial evaluation. Those subjects agreeing to enter the study will have portions of the blood, urine and CSF preserved for study purposes. Study subjects will be followed from the time of hospital admission until death or 1-2 weeks post hospital discharge. Primary study objectives are to: determine whether African children with cerebral malaria (CM) have sufficient levels of systemic tetrahydrobiopterin (BH4) by analyzing their urine for metabolites of BH4; determine whether these children have sufficient levels of BH4 in their CNS by analyzing their cerebrospinal fluid for BH4 metabolites; and determine whether these children have sufficient levels of BH4-dependent biogenic amine neurotransmitters in their CNS by analyzing their cerebrospinal fluid (CSF) for metabolites of the neurotransmitters. Secondary objectives are to: determine natural history of hyperphenylalaninemia in CM and correlate with outcome (i.e., death or recovery); and determine whether BH4 deficiency is due to low expression of genes encoding de novo BH4 synthesis in peripheral blood mononuclear cells from children with CM.

ELIGIBILITY:
Inclusion Criteria:

Uncomplicated malaria (UM) Inclusion Criteria:

* Age between 6 months and 6 years, male and female.
* P. falciparum parasitemia (greater than or equal to 10,000 trophozoites/microliter).
* Clinical syndrome consistent with malaria associated with documented fever (axillary temperature greater than or equal to 38 degrees C) or reported history of fever in the last 48 hours with no other cause present.
* No other infection identified (ie. Negative blood and/or urine cultures).
* Commenced oral quinine less than or equal to 8 hours prior to enrollment.
* Parental permission obtained from parent or legal guardian.

Cerebral Malaria (CM) Inclusion Criteria:

* Age between 6 months to 6 years, male and female.
* Coma (Blantyre Coma Score less than or equal to 2) which persists for > 30 minutes after correction of hypoglycemia and/or seizure.
* Other causes of coma excluded by lumbar puncture.
* Any degree of P. falciparum parasitemia.
* Less than 8 hours since commencement of intravenous quinine (ideally not yet commenced or soon after).
* Parental permission obtained from parent or legal guardian.

Non-malaria CNS disease (NMC) Inclusion Criteria:

* Age between 6 months and 6 years, male and female.
* Non-malaria cause of altered consciousness/coma identified (eg. Meningitis, subarachnoid hemorrhage, trauma, metabolic, toxic, post-ictal febrile seizure).
* Parental permission obtained from parent or legal guardian.

Healthy Control (HC) Inclusion Criteria:

* Age between 6 months and 6 years, male and female.
* No febrile illness within 2 weeks of evaluation.
* No active inflammatory condition identified.
* Parental permission obtained from parent or legal guardian.
* Negative RDT (rapid diagnostic test for malaria).

Exclusion Criteria:

Uncomplicated malaria (UM) Exclusion Criteria:

* Mixed infection with P. falciparum and any other malaria species (P. malariae, P. ovale, P. vivax).
* Co-infection with any other organism identified (ie. Positive blood culture).
* On quinine or artemesinin derivatives for greater than or equal to 8 hours.
* Presence of warning signs suggesting more severe disease, including the following:

  1. Unable to suckle, eat and/or drink
  2. Excessive vomiting
  3. Abnormal respiration/respiratory distress (use of accessory muscles of respiration, tracheal tugging, intercostal retractions)
  4. Recent history of convulsions
  5. Altered mental state
  6. Prostration (unable to sit unaided)

Cerebral Malaria (CM) Exclusion Criteria

* Untreated severe malaria anemia (hemoglobin less than or equal to 6 gm/dl).
* Lumbar puncture not performed.
* Mixed infection with P. falciparum and any other malaria species (P. malariae, P. ovale, P. vivax).
* On quinine or artemesinin derivatives for greater than or equal to 8 hours.

Non-malaria CNS disease (NMC) Exclusion Criteria:

* Lumbar puncture not performed.
* Untreated severe anemia (hemoglobin less than or equal to 6.0 gm/dl due to any cause).
* Any degree of P. falciparum parasitemia.

Healthy Control (HC) Exclusion Criteria

* Fever (Temp > 38.0 degrees C).
* History of sickle cell disease or sickle cell trait.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study is a prospective cohort study involving Tanzanian children 6 months to 6 years old admitted with UM and CM as defined by World Health Organization (WHO) criteria (Section 5.2). Healthy children who are not acutley ill (healthy control, HC) and children with coma and/or CNS illnesses not attributed to malaria (NMC) will serve as controls. Children will be recruited from 2 hospitals in Dar es Salaam (AHID,MDH).
Sampling Method: Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Granger, M.D., Principal Investigator — University of Utah, Division of Infectious Diseases; Esther D. Mwaikambo, M.D., Principal Investigator — Hubert Kairuki Memorial Hospital (HKMU)
Locations (1):
- Hubert Kairuki Memorial University, Dar es Salaam, Tanzania